CLINICAL TRIAL: NCT00877500
Title: A Phase II Randomized Study of Ixabepilone vs. Observation in Patients With Significant Residual Disease After Neoadjuvant Systemic Therapy for HER2/Neu-Negative Breast Cancer
Brief Title: Ixabepilone in Treating Participants With Significant Residual Disease of HER2/Neu Negative Invasive Breast Cancer After Systemic Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0435; NCI-2018-01849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0435 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bilateral Breast Carcinoma; HER2/Neu Negative; Invasive Breast Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; ixabepilone; Epothilones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group I (ixabepilone) (Experimental): Participants receive ixabepilone IV over 3 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ixabepilone
- Group II (standard of care) (Active Comparator): Participants receive standard of care for 18 weeks.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Drug: Ixabepilone — Given IV
  Other Names: (1S,3S,7S,10R,11S,12S,16R)-7,11-Dihydroxy-8,8,10,12,16-pentamethyl-3-[(1E)-1-methyl-2-(2-methyl-4-thiazolyl)ethenyl]-17-oxa-4-azabicyclo[14.1.0]heptadecane-5,9-dione; Azaepothilone B; BMS 247550; BMS-247550; BMS247550; Epothilone; Epothilone-B BMS 247550; Ixempra
  Arms: Group I (ixabepilone)

SUMMARY:
This phase II trial studies how well ixabepilone compared with standard of care works in treating patients with HER2/Neu negative breast cancer that remains after undergoing systemic therapy. Ixabepilone works by blocking cell division which may cause cancer cell death.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the genomic (transcriptional profiles) and proteomic (pathway activation) features that distinguish tumors that do not achieve a pathologic complete response (pCR) after neoadjuvant systemic therapy (NST) and correlate these features with outcome in the presence and absence of adjuvant ixabepilone.

II. To evaluate the presence of circulating tumor cells (CTCs) at baseline (before chemotherapy starts; if radiation is used, after radiation ends), during and after ixabepilone therapy or during observation.

SECONDARY OBJECTIVES:

I. To collect serial blood samples for future pharmacogenomic studies. II. To determine if the addition of adjuvant ixabepilone will improve recurrence-free survival in patients that have significant residual HER 2/neu-negative breast cancer after NST.

III. To assess the toxicity of adjuvant ixabepilone in this group of patients.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I (IXABEPILONE): Participants receive ixabepilone intravenously (IV) over 3 hours on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

GROUP II (STANDARD OF CARE): Participants receive standard of care for 18 weeks.

After completion of study treatment, participants are followed up every 3 months for 2 years and every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic confirmation of invasive HER2/neu-negative breast cancer (immunohistochemistry [IHC] 0-1+ or fluorescence in situ hybridization [FISH]-negative) that have received complete anthracycline and taxane neoadjuvant systemic therapy and that at the time of surgery are expected to have significant residual disease. Therapy should include at least 4 cycles of an anthracycline-based regimen (adriamycin-cytoxan [AC], 5-fluorouracil/adriamycin/intravenous [IV] cyclophosphamide [FAC], fluorouracil-epirubicin-IV cytoxan [FEC]) and 12 weeks of a taxane-based regimen (weekly paclitaxel, every 3-week docetaxel).
* Patients who did not complete therapy due to disease progression are eligible.
* Patients with bilateral breast cancers are eligible.
* Patients should have a Karnofsky performance scale of >= 70%.
* Peripheral granulocyte count of >= 1500/mm^3.
* Platelet count >= 100000 mm^3.
* Bilirubin within normal laboratory values.
* Alkaline phosphatase may be up to 1.5 x upper limit of normal (ULN) of the institution.
* Transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) may be up to 1.5 x upper limit of normal (ULN) of the institution.
* Creatinine levels within normal range.
* Negative serum pregnancy test for a woman of childbearing potential.
* Women of childbearing potential (WOCP) must use a reliable and appropriate contraceptive method during the study and 6 months after chemotherapy is completed. Women of childbearing potential (WOCBP) are women who are not menopausal for 12 months or had no previous surgical sterilization.
* Patients must agree to have study tissue collections and blood sample collections.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with institutional policy.
* Patients should have their surgical tissues evaluated for residual cancer burden (RCB) and be used for correlative studies.
* Sexually active women of childbearing potential must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control.
* All WOCBP MUST have a negative pregnancy test within 7 days prior to first receiving investigational product. If the pregnancy test is positive, the patient must not receive investigational product and must not be enrolled in the study. In addition, all WOCBP will be instructed to contact the Investigator immediately if they suspect they might be pregnant (e.g., missed or late menstrual period) at any time during study participation. The principal investigator (PI) will immediately notify BMS in the event of a confirmed pregnancy in a patient participating in the study.

Exclusion Criteria:

* Patients whose tumors express HER2 protein or have HER2/neu gene amplification.
* Patients with a history of other invasive malignancies diagnosed and treated within the previous 5 years, except non-melanoma skin cancer and non-invasive cervical cancer.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, unstable angina, or congestive heart failure - New York Heart Association Class III or IV, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, chronic liver or renal disease, active upper gastrointestinal [GI] tract ulceration).
* Patients with a pre-existing peripheral neuropathy > grade 1.
* Evidence of distant metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2009-03-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Genomic (transcriptional profiles) and proteomic (pathway activation) features that distinguish tumors | Up to 5 years
  RPPA will be used to objectively quantify (phospho)protein expression. Functional activation of the pathway will be defined as an increase in phosphorylation of at least one half of the components of each pathway above the median RPPA quantified activation across the entire tumor set. Data will be analyzed for the presence of clusters based on differential protein expression by using available methods with the R statistical software package. A variety of unsupervised clustering methods (including hierarchical clustering, K-means, independent component analysis, mutual information, and gene shaving) will be used to classify the samples into statistically similar groups.
Significant circulating tumor cells (CTCs) | At 18 weeks
  Presence of any cell per 7.5 ml of whole blood.

SECONDARY OUTCOMES:
Incidence of adverse events in each group | Up to 5 years
  Chi-square tests of independence and generalized logistic regression models will be used.
Recurrence-free survival | Up to 5 years
  Will be estimated non-parametrically using the Kaplan-Meier product limit method. Cox proportional hazards regression models will be used to model recurrence-free survival as a function of treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Gonzalez-Angulo AM, Lei X, Alvarez RH, Green MC, Murray JL, Valero V, Koenig KB, Ibrahim NK, Litton JK, Nair L, Krishnamurthy S, Hortobagyi GN, Meric-Bernstam F. Phase II Randomized Study of Ixabepilone Versus Observation in Patients With Significant Residual Disease After Neoadjuvant Systemic Therapy for HER2-Negative Breast Cancer. Clin Breast Cancer. 2015 Oct;15(5):325-31. doi: 10.1016/j.clbc.2015.03.004. Epub 2015 Mar 24. PMID 25913905
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org